CLINICAL TRIAL: NCT00167999
Title: Effects of Piperacillin-Tazobactam Use on the Prevalence Rate of Extended-Spectrum Beta-Lactamase (ESBL) Producing Escherichia Coli and Klebsiella Pneumoniae in Hematology and Oncology Units.
Brief Title: Study Evaluating Piperacillin-Tazobactam on Certain Bacteria in Hematology and Oncology Units
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0910X-101676
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Gram-Positive Bacterial Infections; Escherichia Coli Infections; Klebsiella Infections
Keywords: Bacterial Infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Escherichia coli Infections; Klebsiella Infections; Bacterial Infections | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Drug: piperacillin-tazobactam

SUMMARY:
To determine the value of increasing use of piperacillin/tazobactam as empiric therapy and restricting extended-spectrum cephalosporins in reducing the cases of ESBL producing Escherichia coli and Klebsiella pneumoniae in hematology and oncology units

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients of either sex, 15 years of age or older
* Patients who are admitted to the department of hematology and oncology
* Provide written informed consent

Exclusion Criteria:

* Patients who have hypersensitivity to β-lactam antibiotics
* Female who are pregnant or breast-feeding
* Any underlying conditions or non-infectious diseases that will be ultimately fatal within 30 days

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Seoul, South Korea